CLINICAL TRIAL: NCT03657563
Title: An Evaluation of Positive Psychological Intervention on Improving Health of Nurses With Burnout
Brief Title: Improving Health of Nurses With Burnout Through Positive Psychological Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Yuanhui Luo, Principal Investigator, Central South University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2015053
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Nurses with burnout are recruited in the intervention group and participate in positive psychological intervention.
  Interventions: Other: Positive psychological intervention
- Control group (No Intervention): Nurses with burnout are recruited in the control group and none interventions are conducted to them.

INTERVENTIONS:
Other: Positive psychological intervention — Participants in the intervention group are required to record three good things every night before sleeping for five days a week using WeChat. Such things could be ordinary, minor or important.
  WeChat is a common communication tool used in China, just like Facebook, basic messages could be sent individually and posting pictures or texts is also available.
  Arms: Intervention group

SUMMARY:
Burnout is usually regarded as a response to chronic professional stressors like high workload, unfavorable emotion and complex interpersonal relationships. A high prevalence of burnout was found in many countries, and large-scale studies also showed high levels of burnout in Chinese nurses. As a stress-related syndrome, burnout was found to have detrimental influences on both psychological and physical health of nurses. Psychological problems such as depression and insomnia are verified to be associated with burnout. Endocrine dysfunction such as abnormal cortisol secretion rhythm occurred in shift-work nurses. Thyroid dysfunction was increasing and a sample of nurses were diagnosed with thyroid nodules and thyroid hormonal disorder during annual physical examination. Therefore, it is important to take measures to alleviate nurses' burnout to improve health.

Positive psychological interventions are defined as treatment methods or intentional activities to enhance person's positive emotions, cognitions and behaviours. In these methods and activities, people are usually required to finish a systematic exercise. According to a recent meta-analysis, Positive psychological interventions showed effectiveness in enhancing participants' well-being and reducing depressive symptoms. Therefore, this study aims to explore whether positive psychological intervention could reduce burnout and improve health of nurses.

ELIGIBILITY:
Inclusion Criteria:

* officially employed licensed nurses; burnout score higher than 1.49; had a telephone on which WeChat could be installed.

Exclusion Criteria:

* pregnant; current endocrine disorder; taking hormone drugs such as contraceptives.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Burnout at six months | The measurement was taken at baseline and six months.
  Burnout of nurses is measured by Maslach Burnout Inventory-General Survey.
Change from Baseline Morning Plasma Cortisol at six months | The measurement was taken at baseline and six months.
  The level of cortisol is assayed by using chemiluminescence method.
Change from Baseline Thyroid Related Hormones at six months | The measurement was taken at baseline and six months.
  Triiodothyronine (T3), thyroxine (T4) and thyroid stimulating hormone (TSH) are assayed by using chemiluminescence method.

SECONDARY OUTCOMES:
Change from Baseline Resilience at six months | The measurement was taken at baseline and six months.
  Resilience of nurses is measured by Connor-Davidson Resilience Scale.
Change from Baseline Coping at six months | The measurement was taken at baseline and six months.
  The level of coping among nurses is measured by Trait Coping Style Questionnaire.
Change from Baseline Self-efficacy at six months | The measurement was taken at baseline and six months.
  The level of self-efficacy among nurses is measured by General Self-Efficacy Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No